CLINICAL TRIAL: NCT04680572
Title: Functional Outcome After Dual Mobility Cups Total Hip Replacement Versus Bipolar Hemiarthroplasty in Fracture Neck of Femur in Active Elderly Patients
Brief Title: Functional Outcome After Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tony Maher, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD thesis protocol
Record Dates: First submitted 2020-12-13; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Fracture Neck of Femur
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar hemiarthroplasty group (Active Comparator)
  Interventions: Procedure: arthroplasty
- Dual mobility cups total hip replacement group (Active Comparator)
  Interventions: Procedure: arthroplasty

INTERVENTIONS:
Procedure: arthroplasty — arthroplasty for fracture neck of femur

SUMMARY:
Bipolar hemiarthroplasty (BA) has long been the preferred treatment and is performed in most fracture neck of femur (FNF) cases. It is justified by the reasonable operative time, low blood loss and acceptable functional outcomes. The dual mobility cup total hip replacement (DMTHA) has emerged as a relevant alternative to BA. Since then, there is an on-going debate on the best implant to use. Age, co-morbidities, patient independence and potential surgical complications must be considered when deciding between implants. The risk of dislocation is a crucial factor because of its important consequences. The investigators evaluated the functional and mechanical outcomes of BA versus DMTHA in FNF in active elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* active patients
* displaced fracture neck of femur
* age from 60 to 80

Exclusion Criteria:

* ipsilateral previous hip surgery
* grade 3 hip osteoarthritis according to tonnis classifiction
* dysplastic acetabulum

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
functional outcome using the Harris hip score | 2 years
  hip joint range of motion and activities of daily living
rate of dislocation | 2 years
  postoperative prosthesis dislocation

SECONDARY OUTCOMES:
operative time in minutes | 45 minutes to 2 hours
  the time needed to perform the procedure
blood loss in cc | during the procedure
  the amount of blood loss during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim M Ganzoury, professor, Study Director — Faculty of Medicine Ain Shams university
Locations (1):
- Ain Shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
demographic data and radiographs
Supporting Information: Study Protocol, SAP, ICF, CSR

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT04680572/Prot_SAP_000.pdf